CLINICAL TRIAL: NCT07266818
Title: A Multiple Dose Study to Evaluate Safety, Tolerability, PK, and Effect of MK-1167 on QTc in Healthy Adult Participants
Brief Title: A Clinical Trial of MK-1167 in Healthy Adults (MK-1167-010)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1167-010
Record Dates: First submitted 2025-12-01; First posted 2025-12-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-1167 (Experimental): MK-1167 administered orally
  Interventions: Drug: MK-1167
- Placebo (Placebo Comparator): Placebo for MK-1167 administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-1167 — Oral capsule administered once daily
  Arms: MK-1167
Drug: Placebo — Oral capsule administered once daily
  Arms: Placebo

SUMMARY:
The goal of this trial is to learn about the safety of MK-1167 and if people tolerate it.

ELIGIBILITY:
The key inclusion criteria but are not limited to the following:

* Is in good health
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2, inclusive

The key inclusion criteria but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases
* Is a smoker and/or has used nicotine or nicotine-containing products (for example, nicotine patch and electronic cigarette) within the past 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 9 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 1 week
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Hassman Research Institute Marlton Site ( Site 0001), Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com